CLINICAL TRIAL: NCT06160791
Title: Frontline Ruxolitinib With De-Intensified HLH-94 for Adult Hemophagocytic Lymphohistiocytosis (HLH): A Multicenter, Single-Arm Phase 2 Study
Brief Title: Ruxolitinib With De-Intensified HLH-94 for the Treatment of Hemophagocytic Lymphohistiocytosis (HLH)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jerry Lee, MD, MSc, MPhil (Other)
Collaborators: Incyte Corporation (Industry); UC Hematological Malignancies Consortium (UCHMC) (Unknown)
Responsible Party: Sponsor-Investigator, Jerry Lee, MD, MSc, MPhil, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 232513; NCI-2023-09578 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hemophagocytic Lymphohistiocytoses
Keywords: HLH-94
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — ruxolitinib; Janus Kinases; Etoposide; Dexamethasone; Absorptiometry, Photon; High-Energy Shock Waves; Magnetic Resonance Spectroscopy; Biopsy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ruxolitinib, dexamethasone, etoposide) (Experimental): During induction therapy, participants receive ruxolitinib orally (PO) twice daily (BID) plus de-intensified HLH-94 induction with dexamethasone PO or intravenously (IV) once daily (QD) or BID for 4 weeks and etoposide IV twice a week (BIW) for 2 weeks and then based on response, once a week (QW) for another 2 weeks in the absence of disease progression or unacceptable toxicity. After induction therapy, participants receive continuation therapy with ruxolitinib PO BID on days 1-28 of each cycle. Treatment repeats every 28 days for a total of up to 6 months after first administration of study drug in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ruxolitinib; Drug: Etoposide; Drug: Dexamethasone; Procedure: Non-interventional Imaging; Procedure: Research Biopsy; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Ruxolitinib — Administered Orally (PO)
  Other Names: INCB18424; Oral JAK
Drug: Etoposide — Administered IV
  Other Names: Toposar; Lastet
Drug: Dexamethasone — Administered PO or IV
  Other Names: Dexa
Procedure: Non-interventional Imaging — Participants undergo abdominal ultrasound and/or magnetic resonance imaging (MRI)
  Other Names: Ultrasound; Magnetic resonance imaging (MRI)
Procedure: Research Biopsy — Bone marrow biopsy and lymph node biopsy will be obtained during screening and as clinically indicated throughout the trial.
  Other Names: Biopsy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Specimen collection

SUMMARY:
This phase II trial tests the effects of ruxolitinib in combination with a de-intensified HLH-94 drug regimen has on patients with newly diagnosed hemophagocytic lymphohistiocytosis (HLH), a disorder caused by dysregulated immune responses (that is, immune responses that are too strong and cause inflammatory damage to normal tissues). The therapy used for HLH decreases the activity of the immune system. Ruxolitinib is a type of drug called a kinase inhibitor. It works by blocking the signals that cause inflammatory cells to multiply. De-intensified HLH-94 is a treatment regimen that includes 4 weeks of dexamethasone with the dose being decreased each week, and up to 4 weeks of etoposide. This combination is commonly used to treat HLH. Dexamethasone is a steroid medication that works by fighting inflammation. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and deoxyribonucleic acid (DNA) repair and may kill cancer cells and is used to kill the types of white blood cells in HLH that are attacking the body. Giving ruxolitinib in combination with a de-intensified HLH-94 drug regimen may reduce toxic exposure to therapy while maintaining efficacy in patients with HLH.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of ruxolitinib with de-intensified HLH-94 (dHLH-94; 4 weeks of dexamethasone and etoposide) for newly diagnosed adults with HLH.

SECONDARY OBJECTIVES:

I. To describe the toxicities of ruxolitinib in combination with de-intensified HLH-94 for the treatment of adult HLH.

II. To evaluate best response, time to best response, and duration of response stratified by mHLH and nmHLH.

III. To evaluate the progression-free survival (PFS) of using ruxolitinib in combination with dHLH-94 for the treatment of adult HLH, stratified by malignancy-associated hemophagocytic lymphohistiocytosis (mHLH) and non-malignancy-associated hemophagocytic lymphohistiocytosis (nmHLH).

IV. To evaluate the overall survival (OS) when using ruxolitinib in combination with de-intensified HLH-94 for the treatment of adult HLH, stratified by mHLH and nmHLH.

V. To evaluate the time to cancer diagnosis for HLH, among those ultimately diagnosed with mHLH.

VI. To evaluate the time to cancer-directed therapy from the diagnosis of mHLH. VII. To describe the practice patterns of adjunctive therapies (i.e., rituximab, intravenous immunoglobulin therapy (IVIG), anakinra) for HLH.

EXPLORATORY OBJECTIVES:

I. To identify T cell subsets that are differentially increased in adult HLH (comparing mHLH and nmHLH).

II. To evaluate the association of CD8+ T cell subsets expressing CD4dim/CD38+/HLA-DR+ ("activated T cells") with clinical deterioration.

III. To evaluate the relationship between the peripheral blood cytokine microenvironment (e.g., Interleukin 1b (IL-1b), Interleukin 2 (IL-2), Interleukin 6 (IL-6), Interleukin 10 (IL-10), Interleukin 18 (IL-18), Interferon gamma (IFN-gamma), Tumor Necrosis Factor alpha (TNF alpha), laboratory parameters (ferritin, blood counts, liver function, fibrinogen), and response to ruxolitinib.

OUTLINE:

During induction therapy, participants receive ruxolitinib plus de-intensified HLH-94 induction with dexamethasone and etoposide and then based on response, another 2 weeks of treatment will be given in the absence of disease progression or unacceptable toxicity. After induction therapy, participants receive continuation therapy with ruxolitinib for a total of up to 6 months after first administration of study drug in the absence of disease progression or unacceptable toxicity. After completion of study treatment, participants are followed up at 30 days and then at 3, 6, and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Males and females, 18 years of age or older at the time of enrollment.
* Participants must have active HLH and meet >= 5 of 8 of the HLH-2004 diagnostic criteria, or have familial/primary HLH with pathogenic/likely pathogenic germline variant(s) in genes known to cause HLH (e.g., PRF1, UNC13D, Syntaxin 11 (STX11), Syntaxin-binding protein 2 (STXBP2), RAB27A, SH2 domain-containing protein 1A (SH2D1A), baculovirus inhibitor of apoptosis repeat containing protein 4 (BIRC4), Lysosomal trafficking regulator (LYST), interleukin-2-inducible T-cell kinase (ITK), SLC7A7, X-linked immunodeficiency with magnesium defect, Epstein-Barr virus infection, and neoplasia (XMEN), Hermansky-Pudlak syndrome (HPS), NLR family CARD domain-containing protein 4 (NLCR4) or other immune regulatory genes.

  * Fever >= 38.5 degrees Celsius (C) (or >= 38 degrees C if acetaminophen given in prior 6 hours).
  * Splenomegaly.
  * Peripheral cytopenias involving >= 2 of 3 cell lines (absolute neutrophil count < 1000/uL; hemoglobin < 9 g/dL; platelets < 100,000/uL).
  * Hypertriglyceridemia (fasting triglycerides >= 265 mg/dL) or Hypofibrinogenemia (fibrinogen =< 150 g/dL).
  * Hemophagocytosis on tissue biopsy, such as in the bone marrow, spleen, lymph node, or liver.
  * Low/absent natural killer (NK)-cell activity/perforin and/or decreased CD107a mobilization.
  * Ferritin >= 500 ug/L.
  * Soluble IL-2 receptor (sCD25) > 2400 U/mL or two standard deviations above age-adjusted laboratory-specific norms.
* The effects of ruxolitinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception for the duration of study participation and for two months after last administration of study treatment.

  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and two months after last administration of study treatment.

Exclusion Criteria:

* Participant is receiving or received any other investigational agent within 1 week of the first dose of treatment.
* Females who are pregnant or breastfeeding. Female participants of child-bearing potential must have a negative pregnancy test within 7 days of treatment and lactating females must discontinue breast feeding during treatment and until two weeks after the final dose of ruxolitinib.
* Males who expect to conceive children, and/or who decline highly effective methods of contraception during the entire duration of the study.
* Patient cannot take medications orally or via a nasogastric/orogastric tube.
* Poor life expectancy < 2 weeks.
* Clinically significant or uncontrolled cardiovascular disease, including unstable angina, acute myocardial infarction, or stroke within 6 months, New York Heart Association class III or IV. congestive heart failure, and arrhythmia requiring therapy or uncontrolled hypertension (blood pressure > 170/100 mmHg) unless approved by the sponsor- investigator.
* Estimated creatine clearance (CrCl) < 15 mL/min while not on dialysis.
* Known (biopsy-confirmed) liver cirrhosis or suspected cirrhosis with a Model for End- Stage Liver Disease (MELD) score of > 20, or aspartate aminotransferase (AST) or alanine transaminase (ALT) values > 1000 not expected to improve with HLH therapy.
* Severe organ dysfunction, such as cardiorespiratory failure requiring inotropic medications or extracorporeal life support. Respiratory support including intubation/ventilation is allowed.

  * Vasopressors are allowed if not required other than low dose vasoconstrictors to compensate the effects of sedation.
* Newly diagnosed acute and clinically active tuberculosis, hepatitis B, and/or hepatitis C.

  * Patients with active human immunodeficiency virus (HIV) are not excluded from this study but must be on antiretrovirals.
  * Patients with hepatitis B or C viremia can be on study if the hepatitis is not considered clinically active and/or if it is chronic. These patients should be discussed with the principal investigator.
* Individuals with a prior malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Individuals with chimeric antigen receptor (CAR)-T-associated HLH.
* No prior HLH-directed therapy except corticosteroids for < 2 consecutive weeks and anakinra.

  * Adjunctive approaches such as rituximab for Epstein-Barr virus (EBV) viremia or IVIG for viral infection are permitted.
  * Emapalumab, alemtuzumab, anti-thymocyte globulin (ATG), tocilizumab, siltuximab, or prior ruxolitinib are NOT permitted. Cyclosporine and tacrolimus are not permitted in the initial induction period.
* Hypersensitivity to ruxolitinib or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 4 weeks
  The proportion of responder (complete response (CR), complete response with incomplete hematologic recovery, or partial response (PR)) or non-responder at the end of induction using a physician developed response criteria will be reported. Those with non-malignant HLH (nmHLH) will be assessed for response, defined as complete response (CR) + partial response (PR) at 4 weeks. Participants diagnosed with a malignant trigger are recommended to undergo cancer-directed therapy once acute hypercytokinemia improves. The primary endpoint for malignant HLH (mHLH) is achievement of PR or better and initiation of cancer-directed therapy (non-HLH specific therapy) by 4 weeks.

SECONDARY OUTCOMES:
Proportion of participants reporting high-grade adverse events | Up to 1 year
  Safety analyses will be descriptive and performed based on the safety population, defined as patients who received at least one dose of study drug. Serious adverse events (SAEs), adverse events (AEs) ≥ grade 3, and AEs resulting in discontinuation of treatment, withdrawal from the study, and deaths on-study will be tabulated.
Best Response Rate | Up to 1 year
  The proportion of responders by best response defined as a complete response (CR), complete response with incomplete hematologic recovery, partial response (PR) or stable disease (SD)) using a physician developed response criteria will be reported.
Median Time to Best Response | Up to 12 months after the end of continuation therapy, approximately 2 years total
  The median time in months from the time of treatment initiation until participants best response at 12 months after the end of continuation therapy will be reported.
Median Duration of Best Response | Up to 12 months after the end of continuation therapy, approximately 2 years total
  The median time in months from the participants obtained a best response from until 12 months after the end of continuation therapy, participant withdrawal, or death will be reported.
Median progression free survival (PFS) | Up to 1 year
  PFS is defined as the median number of months from first dose to disease relapse, progression, or death, whichever occurs first using using Kaplan-Meier methods.
Median overall survival (OS) | Up to 1 year
  OS is defined as the median number of months from first dose to until death or study discontinuation, whichever occurs first using using Kaplan-Meier methods.
Median time from the diagnosis of hemophagocytic lymphohistiocytosis (HLH) to diagnosis of cancer | Up to 1 year
  The duration of time in days from the diagnosis of hemophagocytic lymphohistiocytosis (HLH) to the diagnosis of cancer will be reported.
Median time from diagnosis of malignancy-associated HLH to initiation of cancer-directed therapy | Up to 1 year
  The duration of time in days from the diagnosis of malignancy-associated hemophagocytic lymphohistiocytosis to the initiation of cancer-directed therapy will be reported using Kaplan-Meier methods.
Number of different adjunctive therapies | Up to 2 years
  The number of adjunctive therapies for HLH will be reported by type, frequency, and indication.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Lee, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with study collaborators during the course of the study.
Supporting Information: Study Protocol, SAP